CLINICAL TRIAL: NCT04043208
Title: Tratamiento de la Distension Abdominal Funcional
Brief Title: Treatment of Functional Abdominal Distension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)377/2018
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Irritable Bowel Syndrome; Dyspepsia
MeSH Terms: conditions — Irritable Bowel Syndrome; Dyspepsia | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental)
  Interventions: Behavioral: Biofeedback
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Biofeedback — Three sessions of biofeedback will be performed during the first 3 weeks of the intervention period. Biofeedback sessions will be performed 30 min after ingestion of the offending meal: patients will be taught to control abdominal and thoracic muscular activity by providing a visual display of the abdominal and thoracic perimeter; specifically, they will be instructed to reduce the abdominal perimeter (girth). Patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period.
  Arms: Biofeedback
Dietary Supplement: Placebo — Three sessions will be performed during the first 3 weeks of the intervention period. Each session will be performed 30 min after ingestion of the offending meal: abdominal and thoracic perimeter will be recorded but not shown to the patient; patients will take a pill of placebo containing 0.5 g glucose and no specific instructions will be provided. Patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.
  Arms: Placebo

SUMMARY:
Background. Abdominal distention is produced by an abnormal somatic postural tone. We developed an original biofeedback technique based on electromyography-guided control of abdominothoracic muscular activity. In a randomized, placebo-controlled trial we demonstrated the superiority of biofeedback over placebo for the treatment of abdominal distention. However, the technique is technically complex and unpractical.

Aim. To prove the efficacy of a simplified biofeedback technique for the treatment of abdominal distension.

Selection criteria. Visible abdominal distension after meal ingestion; patients are able to identify the offending meal.

Intervention. Patients will be randomized into biofeedback in placebo groups.Three sessions of either biofeedback or placebo intervention will be performed 30 min after ingestion of the offending meal during the first 3 weeks of the intervention period.

Biofeedback: patients will be taught to control abdominal and thoracic muscular activity by providing a visual display of the abdominal and thoracic perimeter; specifically, they will be instructed to reduce the abdominal perimeter (girth); patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period.

Placebo: abdominal and thoracic perimeter will be recorded but not shown to the patient and a pill of placebo containing 0.5 g glucose will be administered; patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.

Primary Outcome Measure:

Effect of the probe meal on the activity of thoraco-abdominal muscles (intercostals, external oblique, internal oblique, upper rectus, lower rectus) measured by electromyography before and after the probe meal. The response to the probe meal will be measured before and after treatment.

Secondary Outcome Measures:

* Effect of the probe meal on sensation of abdominal distension measured by 0-6 scales after the probe meal.
* Changes in girth produced by the probe meal measured using a non-stretch belt placed over the umbilicus before and after the probe meal.
* Sensation of abdominal distension measured by 0-6 scales after each meal (breakfast, lunch, dinner) over a 7-day clinical evaluation period before and during the 4th week of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* episodes of visible abdominal distension triggered by meal ingestion
* patients are able to identify the offending foodstuff

Exclusion Criteria:

* organic cause detected by clinical work-up
* constipation
* abdominal distension not confirmed by the 7-day clinical questionnaires of after the probe meal in the pre-intervention evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Effect of the probe meal on thoraco-abdominal activity of the muscular walls. | 4 weeks
  Activity of thoraco-abdominal muscles (intercostals, external oblique, internal oblique, upper rectus, lower rectus) will be measured by electromyography before and after the probe meal. The response to the meal will be measured before and after treatment.

SECONDARY OUTCOMES:
Effect of the probe meal on sensation of abdominal distension | 4 weeks
  Sensation score measured by 0-6 scales after the probe meal.The response to the meal will be measured before and after treatment.
Changes in girth produced by the probe meal | 4 weeks
  Abdominal girth will be measured using a non-stretch belt that is placed over the umbilicus before and after the probe meal.The response to the meal will be measured before and after treatment.
Sensation of abdominal distension | 4 weeks
  Sensation score measured by 0-6 scales after each meal (breakfast, lunch, dinner) over a 7-day clinical evaluation period before and during the 4th week of the intervention.
Follow-up after biofeedback | 6 months
  Sensation of abdominal distension measured by 0-6 scales after each meal (breakfast, lunch, dinner) over a 7-day clinical evaluation period at 1, 3 and 6 months after biofeedback treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Barba E, Accarino A, Azpiroz F. Correction of Abdominal Distention by Biofeedback-Guided Control of Abdominothoracic Muscular Activity in a Randomized, Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1922-1929. doi: 10.1016/j.cgh.2017.06.052. Epub 2017 Jul 11. PMID 28705783
- [Derived] Barba E, Livovsky DM, Accarino A, Azpiroz F. Thoracoabdominal Wall Motion-Guided Biofeedback Treatment of Abdominal Distention: A Randomized Placebo-Controlled Trial. Gastroenterology. 2024 Aug;167(3):538-546.e1. doi: 10.1053/j.gastro.2024.03.005. Epub 2024 Mar 11. PMID 38467383